CLINICAL TRIAL: NCT01442649
Title: Phase II, Multicentric Randomized Trial, Evaluating the Efficacy of Fluoropyrimidine-based Standard Chemotherapy, Associated to Either Cetuximab or Bevacizumab, in KRAS Wild-type Metastatic Colorectal Cancer Patients With Progressive Disease After Receiving First-line Treatment With Bevacizumab
Brief Title: Efficacy of Chemotherapy, Associated to Either Cetuximab or Bevacizumab, in KRAS Wild-type Metastatic Colorectal Cancer Patients With Progressive Disease After Receiving First-line Treatment With Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 18 / ACCORD 22/0906
Record Dates: First submitted 2011-09-05; First posted 2011-09-28 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer
Keywords: Adenocarcinoma; Metastatic; Second-line treatment; Progressive disease after first-line treatment with bevacizumab; Non-mutated (wild-type) KRAS.
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Oxaliplatin; Leucovorin; Irinotecan; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : bevacizumab + fluoropyrimidine-based chemotherapy (Experimental): Every 2 weeks :
  - mFOLFOX6 : Oxaliplatin 85 mg/m2 over 120 mn IV on D1, Folinic Acide 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1, 5-fluoro-uracil 400 mg/m² in bolus IV on D1 and 5-fluoro-uracil 2400 mg/m² in infusion IV over 46 h.
  OR
  - FOLFIRI : Irinotecan 180 mg/m2 en 90 mn IV on day D1, Folinic acid 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1, 5-fluoro-uracil 400 mg/m² in bolus IV on D1 and 5-fluoro-uracil 2400 mg/m² in infusion IV over 46 h.
  AND
  Bevacizumab 5 mg/kg IV every 2 weeks.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluoro-uracil; Drug: Irinotecan; Drug: Bevacizumab
- Arm B : cetuximab + fluoropyrimidine-based chemotherapy (Experimental): Every 2 weeks :
  - mFOLFOX6 : Oxaliplatin 85 mg/m2 over 120 mn IV on D1, Folinic Acide 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1, 5-fluoro-uracil 400 mg/m² in bolus IV on D1 and 5-fluoro-uracil 2400 mg/m² in infusion IV over 46 h.
  OR
  - FOLFIRI : Irinotecan 180 mg/m2 en 90 mn IV on day D1, Folinic acid 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1, 5-fluoro-uracil 400 mg/m² in bolus IV on D1 and 5-fluoro-uracil 2400 mg/m² in infusion IV over 46 h.
  AND
  Cetuximab : 500 mg/m² IV every 2 weeks
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluoro-uracil; Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Drug: Oxaliplatin — 85mg/m² over 120 mn on D1 every 2 weeks up to progression or toxicity
Drug: Folinic Acid — 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1 (in the same time that oxaliplatin or irinotecan) every 2 weeks up to progression or toxicity
Drug: 5-fluoro-uracil — 400mg/m² in bolus on D1, then 2400mg/m² over 46 h every 2 weeks up to progression or toxicity
Drug: Irinotecan — 180 mg/m2 over 90 mn IV on D1 every 2 weeks up to progression or toxicity
Drug: Bevacizumab — 5 mg/kg IV over 90 mn on D1 every 2 weeks up to progression or toxicity
  Arms: Arm A : bevacizumab + fluoropyrimidine-based chemotherapy
Drug: Cetuximab — 500mg/m² on D1 every 2 weeks up to progression or toxicity
  Arms: Arm B : cetuximab + fluoropyrimidine-based chemotherapy

SUMMARY:
The main objective is to evaluate progression-free survival (PFS) at 4 months.

The secondary objectives are to evaluate the objective response rate (OR) (= complete responses (CR) and partial responses (PR)) according to the RECIST v1.1 criteria, the progression-free survival (PFS), the overall survival (OS), the overall survival from the date of the first-line chemotherapy used on the metastatic disease, the treatment tolerance (NCI CTC AE V4 criteria, except for peripheral neurological toxicity (Lévi Scale)), the quality of life according to the EORTC QLQ-C30 criteria.

The objectives of the biological study are to evaluate potentially predictive anti-EGFR and anti-VEGF response factors and CEC rates as predictive biomarkers for the efficacy of bevacizumab associated with chemotherapy in mCRC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon expressing non-mutated (wild-type) KRAS.
* Progressive metastatic disease after first-line treatment with chemotherapy alone: based on 5-FU (iv or per os) with irinotecan or oxaliplatin associated to bevacizumab.
* Prior adjuvant chemotherapy (of the primary tumor) with fluoropyrimidine and oxaliplatin is allowed if the time interval between the end of this chemotherapy and the beginning of the first-line metastatic treatment is ≥ 6 months.
* Measurable disease (at least one measurable metastatic lesion) according to the RECIST V1.1 criteria (the lesion should not be located in a previous field of radiation).
* Previous radiotherapy is authorized if discontinued ≥ 15 days prior to randomization and if the measurable metastatic lesions are outside the radiation area.
* Sites of disease evaluated within 28 days prior to randomization with thoracic-abdominal-pelvic CT scan (or abdominal-pelvic MRI plus Chest Xray)
* Age ≥18 years
* Patient with ECOG 0 or 1
* Life Expectancy ≥ 3 months
* Hematologic function (polynuclear neutrophiles ≥ 1.5.109/L ; platelets ≥ 100.109/L ; hemoglobin ≥ 9 g/dL
* Hepatic transaminases ≤ 2.5 times upper limit of normal (ULN) (≤ 5 ULN in case of hepatic metastases), alkaline phosphatases ≤ 2.5 ULN (≤ 5 ULN in case of hepatic metastases), total bilirubinemia ≤ 1.5 ULN
* Renal function (creatinemia ≤1.5 ULN; creatine clearance ≥ 50 mL/mn (Cockcroft and Gault) ; urine test strip < 2+. If proteinuria is ≥ +2 at inclusion, the serum urea test must be redone and show proteinuria ≤ 1 g/L within 24 h)
* Completion of the EORTC QLQ-C30 quality of life form
* Negative pregnancy test for women of child-bearing age
* Information given to the patient and signed informed consent
* Public Health insurance coverage

Exclusion Criteria:

* Known meningeal or brain metastases
* Pre-treatment with anti-EGFR
* Specific contraindication or known hypersensitivity to one treatment product
* Patient with known allergy or hypersensitivity to monoclonal antibodies (bevacizumab, cetuximab
* Clinically significant affection of the coronaries or myocardial infarction within 6 months prior to inclusion.
* Peripheral neuropathy of grade > 1 (CTCAE scale version 4.0).
* Known depletion of the dihydropyrimidine dehydrogenase (DPD).
* Acute intestinal obstruction or sub-obstruction, history of inflammatory intestinal disease or extended resection of the small intestine. Presence of a colic prosthesis.
* Uncontrolled Arterial hypertension (systolic pressure > 150 mmHg and/or diastolic pressure > 100 mmHg with and without antihypertensive medication. Patients with high hypertension are eligible if antihypertensive medication lowers their arterial pressure to the level of acceptability specified by the inclusion criteria.
* History of hypertensive crisis or hypertensive encephalopathy
* Other concomitant malignancy or history cancer (except carcinoma in situ of the cervix, or non melanoma skin cancer, with curative intent treatment, when considered in complete remission for at least 5 years before randomization.
* Any treatment including an experimental drug, or participation in another clinical trial within 28 days preceding inclusion.
* Persons deprived of liberty or under guardianship.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 4 months | 4 months
  Progression-free survival is defined as the time from randomization to progression (RECIST v1.1 criteria) or death. Patients alive without progression will be censored at the last follow-up.

SECONDARY OUTCOMES:
Objective response rate (OR) | 12 months
  The objective response rate is defined as the occurence of a complete response [CR] or a partial responses [PR] according to RECIST V1.1 between date of randomization and date of end of treatment. It will be evaluated by the investigator with RECIST v1.1 criteria every 6 weeks up to disease progression.
Progression-free survival (PFS) | 4 months
  Progression-free survival is defined as the time from randomization to progression (RECIST v1.1 criteria) or death. Patients alive without progression will be censored at the last follow-up.
Overall survival (OS) | until death or progression (24 months)
  Overall survival is defined as the time from randomization to death any cause or last follow-up (censored data).
Overall survival from the date of the first-line chemotherapy used on the metastatic disease | until death or progression (24 months)
  Overall survival from the date of the first-line chemotherapy used on the metastatic disease is defined as the time from the first day of the first-line chemotherapy used on the metastatic disease to death any cause or last follow-up news (censored data).
Treatment tolerance | Every 2 weeks, during the treatment.
  Tolerance of the treatment will be based on toxicities of evaluated products by clinical and biological measurements (NCIC/CTC (CTCAE V4) criteria, except for peripheral neuropathy toxicity (Lévi scale)).
Quality of life | every 6 weeks
  Quality of life will be evaluated with the EORTC QLQ - C30.

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, Dr, Principal Investigator — Centre René Gauducheau; Christophe BORG, Pr, Principal Investigator — CHU Jean Minjoz-BESANCON; Christian BOREL, Dr, Principal Investigator — Centre Paul Strauss-STRASBOURG; Jean-Pierre DELORD, Pr, Principal Investigator — Institut Claudius Regaud-TOULOUSE; Christophe BORG, Pr., Principal Investigator — Centre Hospitalier du Mittan-MONTBELIARD; Jean-François SEITZ, Pr, Principal Investigator — CHU Timone-MARSEILLE; Thierry CONROY, Pr, Principal Investigator — Centre Alexis Vautrin-VANDOEUVRE LES NANCY; Roger FAROUX, Dr, Principal Investigator — CHD Vendée-LA ROCHE SUR YON; Eric FRANCOIS, Dr, Principal Investigator — Centre Antoine Lacassagne, Nice; Alice GAGNAIRE, Dr, Principal Investigator — Hôpital Bocage-DIJON; Antoine ADENIS, Pr, Principal Investigator — Centre Oscar Lambret-LILLE; Cédric LECAILLE, Dr, Principal Investigator — Polyclinique Bordeaux Nord Aquitaine-BORDEAUX; Gaël DEPLANQUE, Dr, Principal Investigator — Groupe hospitalier St Joseph-PARIS; Pascal ARTRU, Dr, Principal Investigator — Hôpital Privé Jean Mermoz-LYON; Oana COJOCARASU, Dr, Principal Investigator — Centre hospitalier du Mans-LE MANS; Laurent MIGLIANICO, Dr, Principal Investigator — CHP Saint Grégoire-SAINT GREGOIRE; Olivier BOUCHE, Pr, Principal Investigator — Hôpital Robert Debré - CHU Reims; You-Heng LAM, Dr, Principal Investigator — Centre Hospitalier de Cholet; David TOUGERON, Dr, Principal Investigator — CHU de Poitiers-POITIERS; Barbara DAUVOIS, Dr, Principal Investigator — CHR d'Orléans - Hôpital la Source; Philippe HOUYAU, Dr, Principal Investigator — Clinique Claude Bernard, Albi
Locations (1):
- Centre rené Gauducheau, Saint-Herblain, France

REFERENCES:
- [Derived] Bennouna J, Hiret S, Bertaut A, Bouche O, Deplanque G, Borel C, Francois E, Conroy T, Ghiringhelli F, des Guetz G, Seitz JF, Artru P, Hebbar M, Stanbury T, Denis MG, Adenis A, Borg C. Continuation of Bevacizumab vs Cetuximab Plus Chemotherapy After First Progression in KRAS Wild-Type Metastatic Colorectal Cancer: The UNICANCER PRODIGE18 Randomized Clinical Trial. JAMA Oncol. 2019 Jan 1;5(1):83-90. doi: 10.1001/jamaoncol.2018.4465. PMID 30422156